CLINICAL TRIAL: NCT03373981
Title: Non-invasive Brain Stimulation for the Treatment of Depression Symptoms in ALS: A Pilot Study
Brief Title: Non-invasive Brain Stimulation for the Treatment of Depression Symptoms in ALS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not meet target enrollment
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0326
Record Dates: First submitted 2017-11-30; First posted 2017-12-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: ALS

STUDY DESIGN:
Intervention Model Description: open label single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- intervention (Experimental): rTMS
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — repetitive transcranial magnetic stimulation

SUMMARY:
This is an open-label clinical trial to determine the safety of rTMS and efficacy in improving depression symptoms, quality of life and cognition deficits among patients with Amyotrophic Lateral Sclerosis (ALS) and other neurodegenerative disorders.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the role of repetitive transcranial magnetic stimulation (rTMS) for symptom reduction of depression and cognitive loss among patients with Amyotrophic Lateral Sclerosis (ALS) and other Neurodegenerative Diseases. Behavioral symptoms in ALS have been under scrutiny since its earliest descriptions, nearly 30 years ago (1). The importance of these symptoms among subjects with ALS has been also been under steady scrutiny. Studies have shown that the rates of anxiety and depression are significantly higher among subjects with ALS than the general population (1-23). Anxiety symptoms are related to depression, quality of life, and satisfaction with life (4, 9, 11, 15, 20, 24-26). Depressive symptoms are closely related to the ALS disease process (2).

rTMS has been shown to be a promising tool in modulating mood, memory, and cognitive performance (27). Current approaches to the management of ALS involve addressing symptomatology associated with the disease process. Among patients with ALS and other similar Neurodegenerative disorders, it is therefore important to understand if rTMS as an intervention is capable of:

1. Symptomatic improvement in mood,
2. Causing a significant positive change in disease progression or
3. Helping improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of familial or sporadic ALS as well as other Neurodegenerative disorders. Verification of the diagnosis will be performed by the Principal Investigator. This diagnosis can include neuro-degenerative disorders of uncertain cause, including ALS, MND, Peripheral neuropathies, Parkinson's and other progressive motor system diseases.
2. If subjects has ALS diagnosis, the date of dx should be ≤ 2 years
3. Age 18 or older.
4. Capable of providing informed consent.
5. Minimal speech impairment.
6. Ability to comply with study procedures.
7. Ability to communicate clearly if the subject wants to withdraw from the procedure at any stage.
8. MMSE ≥20
9. Female subjects of child bearing potential must engage in abstinence for the duration of the study. If a participant becomes sexually active, she must agree to using the following birth control methods:

   1. Hormonal (oral, implanted, injected, etc)
   2. Intrauterine device in place for ≥ 3 months
   3. Adequate barrier method in conjunction with spermicide
   4. Other
10. Absence of exclusion criteria.

EExclusion Criteria

1. Unable to provide informed consent
2. Significant speech impairment
3. Inability to comply with the procedures
4. Subjects with ALS diagnosis ≥ 2 years
5. Inability to communicate clearly if the subject wants to withdraw from the procedure at any stage
6. Seizures or history of seizures
7. Patients who have underwent brain surgery for any indication
8. Patients with pacemakers, cochlear implants, brain stimulators, infusion pumps, intracardiac lines, metallic clips, other implanted electronic or ferroelectric metallic devices. Dental implants are permitted
9. Inability to perform either TMS or NCS studies due to insufficient MEP or CMAP amplitude.
10. Patients with uncontrolled hypertension
11. Patients with neuro endocrine disorders
12. Patients who are withdrawn from the following drugs within 6 months:

    * Barbiturates
    * Benzodiazepines
    * Meprobamate
    * Chloral hydrate

Patients who have a recent history (within 24h) or chronic history of intake of:

* Cocaine.
* Phencyclidine Phosphate.
* Gamma-Hydroxy Butyrate.
* Amphetamines including N-methylamphetamine, 3,4-Methylenedioxymethamphetamine, 2,5-dimethoxy-4-methylamphetamine, Ephedrine, Cathinone.

  12. Substance abuse+ 13. Excessive use of alcohol # 14. MMSE ≤19 15. Female patients of child bearing potential not practicing contraception 16. Female patients who are pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and efficacy of repetitive transcranial magnetic stimulation (rTMS) using the FDA approved protocol in research subjects with ALS and other Neurodegenerative disorders. | over 4 weeks, done once a week
  Transcranial magnetic stimulation (TMS) is a non-invasive procedure used to stimulate small regions of the brain. It is a FDA approved for treatment resistant depression (K061053). We hypothesize that stimulation of dorsolateral prefrontal cortex (DLPFC) will be safe and effective in patients with ALS and other Neurodegenerative disorders. We will follow the FDA rTMS guidance for industry guidelines. All adverse events from all 15 patients enrolled in the study as assessed by the CTCAE v4.0, and as well, any occurrence of any new seizure in 2 or more patients, as reviewed and assessed by PI and medical monitor.

SECONDARY OUTCOMES:
To understand the impact of rTMS in addressing the mood symptoms associated with ALS. | recorded once a week for the 4 week duration of the study.
  rTMS is known to ameliorate depressive symptoms in patients with treatment resistant depression. It may also ameliorate depressive symptoms in subjects with ALS. This is measured using MQOL (Montreal Quality of life scale). This is a patient-reported instrument designed to assess overall well-being over a two day time scale. this single item scale is scored from 0-10 with higher score representing higher quality of life ratings. percent change from baseline to study completion will be measured to assess the efficacy of rtms in improving overall quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Shara Holzberg, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided